CLINICAL TRIAL: NCT03577613
Title: Radical Hysterectomy: Evolution Of Surgical Approach and Related Outcomes
Acronym: RESurg
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AMI)23/1999
Record Dates: First submitted 2018-05-15; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Surgery--Complications
Keywords: radical hysterectomy; minimally invasive surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early stage Cervical Cancer- Open Radical Hysterectomy(RH): Patients who were clinically diagnosed with FIGO stage IA2-IB1-IIA1 cervical cancer and underwent a open RH at our institution as primary treatment were included in the study
  Interventions: Procedure: Open radical hysterectomy
- Early stage Cervical Cancer- Laparoscopic Radical Hysterectomy: Patients who were clinically diagnosed with FIGO stage IA2-IB1-IIA1 cervical cancer and underwent a laparoscopic RH at our institution as primary treatment were included in the study
  Interventions: Procedure: laparoscopic radical hysterectomy
- Early stage Cervical Cancer- Robotic radical Hysterectomy(RRH): Patients who were clinically diagnosed with FIGO stage IA2-IB1-IIA1 cervical cancer and underwent a robotically assisted RH at our institution as primary treatment were included in the study
  Interventions: Procedure: Robotically assisted radical hysterectomy

INTERVENTIONS:
Procedure: Open radical hysterectomy
  Groups: Early stage Cervical Cancer- Open Radical Hysterectomy(RH)
Procedure: laparoscopic radical hysterectomy
  Groups: Early stage Cervical Cancer- Laparoscopic Radical Hysterectomy
Procedure: Robotically assisted radical hysterectomy
  Groups: Early stage Cervical Cancer- Robotic radical Hysterectomy(RRH)

SUMMARY:
Prospective controlled study (Canadian Task Force II-2) : Comparison analysis regarding surgical outcomes, complications, overall survival (OS), disease free survival (DFS) and cancer specific survival between patients subjected to radical Hysterectomy either by open radical hysterectomy (ORH) or minimally invasive surgery (MIS): laparoscopic (LRH) or robotically assisted radical hysterectomy (RRH).

DETAILED DESCRIPTION:
Study Objective: To analyse the effect that the introduction of minimally invasive procedures has had on surgical and oncological outcomes when compared with conventional open radical hysterectomy (ORH) in a national reference cancer center Design: A prospective controlled study (Canadian Task Force II-2) Setting: A university teaching hospital Patients: All patients that underwent RH as primary treatment for cervical cancer in our institution between May 1999 and June 2016, with a total of 188 patients.

Interventions: Patients underwent an open radical hysterectomy (ORH) or minimally invasive surgery (MIS): laparoscopic (LRH) or robotically assisted radical hysterectomy (RRH).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with FIGO stage IA2-IB1-IIA1 cervical cancer.
* Subjected to Radical Hysterectomy.

Exclusion Criteria:

* Pregnant women in which a RH was performed at the time of caesarean section.
* Previous chemotherapy treatment
* Previous pelvic radiotherapy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients who were clinically diagnosed with FIGO stage IA2-IB1-IIA1 cervical cancer and underwent a RH at our institution
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 1999-05-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Overall survival. | up to 240 months
  From date of randomization until the date of death from any cause.

SECONDARY OUTCOMES:
Disease free survival | up to 240 months
  from surgery to time of recurrence or time of death(all causes)
Cancer specific survival | up to 240 month
  from surgery to time of death( cervical cancer related)
surgical complication Rate | up to 28 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gil-Moreno, MD, PhD, Principal Investigator — Hospital Vall D'Hberon

IPD SHARING:
Plan to Share IPD: Undecided